CLINICAL TRIAL: NCT04492774
Title: GOLDIC Therapy in Lumbar Degenerative Spinal Stenosis - Randomized Controlled Trial
Brief Title: Degenerative Lumbar Stenosis Conservative Treatment
Acronym: GOLDSTEN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sutherland Medical Center (Other)
Responsible Party: Principal Investigator, Piotr Godek, Principal Investigator, Sutherland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC2020002
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Spinal Stenosis Lumbar; Spinal Canal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Dexamethasone; Musculoskeletal Manipulations; Drainage

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Masking Description: None (Open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GOLDIC serum (Experimental): Epidural ultrasound guided injections
  Interventions: Combination Product: Goldic serum
- Steroid (Active Comparator): Epidural ultrasound guided injections
  Interventions: Drug: Steroid injections
- Manual therapy (Active Comparator): veno-lymphatic spinal drainage
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Combination Product: Goldic serum — epidural injections
  Other Names: Autologous serum
  Arms: GOLDIC serum
Drug: Steroid injections — epidural injections
  Other Names: Dexamethasone
  Arms: Steroid
Procedure: Manual therapy — Veno-lymphatic drainage
  Other Names: drainage
  Arms: Manual therapy

SUMMARY:
The trial aims to compare the effectiveness of three methods of conservative treatment of degenerative lumbar spine stenosis (DLSS): GOLDIC autologous serum epidural injections, steroid epidural injections and manual therapy.

DETAILED DESCRIPTION:
BACKGROUND: Degenerative Lumbar Spinal Stenosis (DLSS) is a serious health problem for patients over 65 years of age. It is assumed that in the United States alone, it affects about 200 thousand patients causing significant impairment of their quality of life. Although it is relatively easy to confirm the nature of spinal canal encroaching (disc protrusion, facet hypertrophy, ligamentous folding) by several methods of imaging, the golden standard of DLSS management, especially in the group of older patients, is still the matter of debate. Three main concepts of conservative treatment are considered: 1) pharmacological care - symptom-oriented systemic anty-inflammatory and analgesic agents or local steroid injections, 2) rehabilitations protocols and mechanical devices like traction facilities or corsets to decompress spinal canal or support in case of instability, 3) biological - stimulation of anti-inflammatory action and regeneration capacity by biologically active substances. All methods are offered without strong evidence of its efficacy.

AIM: Comparison of the effectiveness of three treatment protocols in DLSS: epidural injections of autologous serum (Gold Induced Cytokines, Goldic), epidural steroid injections, manual therapy in the concept of spinal canal venous drainage.

Research hypothesis: The use of Goldic serum in epidural injections improves the condition of patients with DLSS during the observation period longer than steroid injections and the rehabilitation protocol.

DESIGN: Randomized prospective trial without blinding. SETTING: Open study for outpatients, single-centre study. POPULATION: the local adult population METHODS: Three groups of patients (A, B, C) with confirmed DLSS in MRI, without limiting sex, age, meeting health conditions according to the inclusion and exclusion criteria. There will be 30 people in each group (90 people in total).

Group A - Goldic serum therapy - 4 injections at 3-day intervals containing single doses of serum (4 doses of 3 ml in total), injections performed into the epidural space under ultrasound control by the same operator.

Group B - steroid therapy with Dexaven 4 mg / 1 ml - 2 injections at weekly intervals containing single doses of dexamethasone (total dose of 8 mg), injections will be performed into the epidural space under ultrasound control by the same operator.

Group C - manual therapy according to the concept of venous drainage - a repeatable treatment scheme for each patient; decompression of the thoracic outlet, diaphragm release, sacroiliac joints (SI) mobilizations, rib-sternum release, rib raising technique - 4 sessions (1 x weekly - approx. 40 min).

Control tools: NRS Pain Scale (0-10), Oswestry Disability Index, Zurich Claudication Questionnaire (ZCQ), EQ-5D-5L, Control points: Initial Assessment (IA), 4,12, 24 weeks after last intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs of lumbar spinal stenosis
2. Radiological signs of lumbar spinal stenosis confirmed by MRI
3. No contraindications to steroid therapy or spinal epidural injections (glaucoma, high RR values, diabetes, anticoagulants, active infections, etc.)
4. Mental state allowing cooperation during manual therapy
5. An adult who consents to participate in the study
6. No previous surgery or spinal epidural injections

Exclusion Criteria:

1. The presence of serious neurological deficits
2. Stenosis of other origin - post-traumatic, spondylolisthesis, cancer, infection
3. Contraindications to steroid therapy or spinal injections (glaucoma, high RR values, diabetes, anticoagulants, active infections, etc.)
4. Previous surgery or spinal epidural injections of lumbar spine
5. Mental state preventing cooperation during manual therapy
6. Lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in EQ-5D-5L index from baseline to 24 weeks | Change from baseline to 24 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
Change in Oswestry Disability Index from baseline to 24 weeks | Change from baseline to 24 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Zurich Claudication Questionnaire (ZCQ) from baseline to 24 weeks | Change from baseline to 24 weeks
  Disease-specific questionnaire. Range: 12 (the best score) - 55 (the worst score).

SECONDARY OUTCOMES:
Change in pain intensity according to Numeric Rating Scale | Change from baseline to 4 weeks
  Generic outcome measure. Range: 0 (no pain) - 10 (the worst possible pain).
Change in pain intensity according to Numeric Rating Scale | Change from baseline to 12 weeks
  Generic outcome measure. Range: 0 (no pain) - 10 (the worst possible pain).
Change in pain intensity according to Numeric Rating Scale | Change from baseline to 24 weeks
  Generic outcome measure. Range: 0 (no pain) - 10 (the worst possible pain).
Change in EQ-5D-5L index from baseline to 4 weeks | Change from baseline to 4 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
Change in EQ-5D-5L index from baseline to 12 weeks | Change from baseline to 12 weeks
  EQ-5D-5L index estimated from EQ-5D-5L desrcriptive system based on Polish directly measured value set. Mininmum: -0.590; Maximum: 1.0; More points means better outcome.
Change in Oswestry Disability Index from baseline to 4 weeks | Change from baseline to 4 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Oswestry Disability Index from baseline to 12 weeks | Change from baseline to 12 weeks
  Disease-specific questionnaire. Range: 0 (the best score) - 50 (the worst score).
Change in Zurich Claudication Questionnaire (ZCQ) from baseline to 4 weeks | Change from baseline to 4 weeks
  Disease-specific questionnaire. Range: 12 (the best score) - 55 (the worst score).
Change in Zurich Claudication Questionnaire (ZCQ) from baseline to 12 weeks | Change from baseline to 12 weeks
  Disease-specific questionnaire. Range: 12 (the best score) - 55 (the worst score).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Godek, PhD, Principal Investigator — Sutherland Medical Center
Locations (1):
- Sutherland Medical Center, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godek P, Szczepanowska-Wolowiec B, Golicki D. GOLDIC therapy in degenerative lumbar spinal stenosis: randomized, controlled trial. Regen Med. 2022 Oct;17(10):709-718. doi: 10.2217/rme-2022-0047. Epub 2022 Jul 28. PMID 35899459